CLINICAL TRIAL: NCT02409277
Title: Redesigning Ambulatory Care Delivery to Enhance Asthma Control in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Flory Nkoy, Associate Professor, University of Utah
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 51002874
Record Dates: First submitted 2015-03-25; First posted 2015-04-06 (Estimated); Results first posted 2020-02-05 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-01

CONDITIONS: Asthma
Keywords: Self-Management; Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant
Masking Description: We initially enrolled 327 randomized (at the clinic level) participants who received the e-AT interventions overall, including 267 participants receiving the standard intervention and 60 receiving the intensive intervention. We also included another set of 599 non-randomized matched controls of patients with persistent asthma retrieved electronically from non-participating clinics. This is why we stated that 926 subjects (327+599) overall were included.
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Standard e-AT Intervention (Experimental): Patients in Standard e-AT or standard intervention group will receive a daily (if a participant forgets to complete his/her weekly assessment) email and text reminders with a link to the e-AT website to help patient/parent participants to comply with their weekly assessment of patient's level of asthma control. Note: patient/parent participants are required to complete their asthma control assessment 1x/week. The e-AT is now set up to send a weekly reminder to participants with a link to the website. If a participant does not complete an assessment within a week of the last assessment, the reminder will be sent daily until the patient/parent complies and the system resets to weekly.
  Interventions: Other: Experimental: Standard vs Intensive e-AT Intervention
- Intensive e-AT Intervention (Experimental): Participants in the intensive e-AT or adherence support intervention will receive everything as those in Standard Intervention. In addition, they will see a progress bar display, which adds 25 points each time they complete an assessment. When this bar reaches 100 points, a pop-up message with fireworks will appear to congratulate them about the milestone. The progress bar resets to zero after it reaches 100 points. Participants will also see a leader board allowing them to compare themselves with the 5 best users to increase compliance.
  Interventions: Other: Experimental: Standard vs Intensive e-AT Intervention
- Usual Care (Non-Randomized Cohort) (No Intervention): Both arms (Intensive and standard e-AT interventions) will be compared to each other as well as to a non-randomized cohort who did not receive the e-AT interventions. These non-randomized cohort will be matched 2:1 to each randomized individuals.

INTERVENTIONS:
Other: Experimental: Standard vs Intensive e-AT Intervention — Patients will be self-monitoring their symptoms weekly using the e-AT, either the Standard or Intensive versions of the e-AT, completing the Asthma Control Test. As patients complete their assessments each week, the clinics will be able to see how each patient is doing, and follow-up when a patient is showing high symptoms for that week, potentially avoiding Emergency Room visit, and/or hospitalization.
  Arms: Intensive e-AT Intervention; Standard e-AT Intervention

SUMMARY:
The investigators have developed a tool to facilitate asthma self-management in children, the electronic-AsthmaTracker (e-AT). The e-AT changes ambulatory asthma care delivery to a new model that is continuous and proactive, focusing on prevention and control, rather than reactive and focusing on management of asthma attacks. The e-AT 1) engages parents in weekly monitoring of their child's chronic asthma symptoms, 2) guides parents to recognize warning signs of asthma attacks in order to prompt appropriate interventions and timely visits to Primary Care Providers, and 3) provides Primary Care Providers with real-time, objective patient data to assess the effectiveness of asthma therapy and prompt adjustments. In a preliminary study of the paper-based version of the AT, frequent users had significantly fewer emergency department (ED) and hospital visits. Parent comments during the e-AT pilot testing revealed that the tool was useful in helping them manage their child's asthma and were interested in assessing the tool's effectiveness and in identifying and addressing barriers to their sustained use of the e-AT.

Improving asthma control in children will be facilitated by broad e-AT dissemination, and by identifying and addressing critical factors that contribute to parent sustained participation in self-management. The investigators propose to assess the effectiveness of the new ambulatory care model supported by the e-AT and conduct an e-AT process evaluation, assessing barriers and facilitators of sustained parent use. The investigators will engage parents throughout this study to identify and address themes that matter to them. The target population is children with persistent asthma, ages 2-17 years. The investigators have engaged 10 parents since conception of this project, from the planning to design and validation of the paper-AT, and the design and pilot testing of the e-AT. Input from parents was received through 3 iterative focus groups (one for the paper-AT and 2 for the e-AT) and facilitated discussions to inform the development of this proposal including research objectives and outcome measures. In addition, the investigators have recruited other key stakeholders for whom the results of the research will be relevant.

DETAILED DESCRIPTION:
Through the following specific aims, the investigators will:

Aim 1: Assess the effectiveness of the new ambulatory care model, by comparing outcomes at the 1.a. child (child's quality of life (QOL), asthma control, missed school days), 1.b.parent (satisfaction, parent missed work days) and 1.c. clinic (ED/hospital visits) levels, between clinics randomly assigned to either the standard e-AT intervention vs. intensive e-AT intervention. 1.d. Use non randomized comparisons to determine the effectiveness of the e-AT relative to a control group (usual care) in which the e-AT was not used

Aim 2: Assess the association of QOL, asthma control, and ED/hospital admissions with the prior frequency of e-AT use and assess if the association differs between parent subgroups (high vs. low literacy, Medicaid vs. private insurance, and frequent vs. less frequent e-AT users).

Aim 3: Determine the association of demographic, socio-economic, behavioral, and technology factors with sustained parent participation in asthma self-management.

The outcome measures are:

Primary Outcome:

1. Child quality of life (QOL)

   Secondary Outcomes:
2. Child asthma control
3. Child interrupted/missed school days
4. Child use of oral steroids (surrogate measure of an asthma exacerbation)
5. Parent satisfaction with care
6. Parent interruption/missed work days
7. Clinics: ED/Hospital admissions

ELIGIBILITY:
Facility Eligibility

Clinics are eligible for participation if they meet the following criteria:

1. Primary care clinics with the clinical leadership to adopt use of e-AT for asthma management.
2. Have patients between 2 and 17 years of age with persistent asthma.
3. Ability of the facility to accommodate patient enrollment and training about use of e-AT.

Patient Inclusion Criteria

1. Children ages 2 through 17 years and their parents (main parents or caregiver)
2. English speakers
3. Children who received or are receiving asthma treatment (at participating clinics).
4. Parents have Internet access
5. Children with persistent asthma.

Patient Exclusion Criteria:

As this is a pragmatic trial assessing evidence of the e-AT in a real clinical environment, no patients will be excluded as long as they meet inclusion criteria. However, during the time of analysis, we will conduct a sub-analysis, comparing the effectiveness of the new care model among patients with or without co-morbid conditions that may affect measured asthma outcomes. These include patients with a history or increased risk of pulmonary disease (cystic fibrosis, bronco-pulmonary dysplasia, aspiration pneumonia, severe Cerebral Palsy (CP) with aspiration risk, technology dependency (gastrostomy tube, tracheostomy), history of congenital heart disease requiring surgical correction or with complicating congestive heart failure requiring medical management, immunodeficiency (including patients on immunosuppressants), and malignancies.

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 926 (Actual)
Dates: Start 2013-08 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Flory Nkoy, MD, MS, MPH, Principal Investigator — University of Utah
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No
We can only share completely de-identified data. Request can be sent to my email: flory.nkoy@hsc.utah.edu

REFERENCES:
- [Background] CDC. National Health Interview Survey (NHIS) Data2009. http://www.cdc.gov/asthma/nhis/09/data.htm
- [Background] Akinbami LJ, Moorman JE, Liu X. Asthma prevalence, health care use, and mortality: United States, 2005-2009. Natl Health Stat Report. 2011 Jan 12;(32):1-14. PMID 21355352
- [Background] CDC. Healthy Youth! Health Topics, Asthma2009.
- [Background] Wessel L, Spain J. The Chronic Care Model: A Collaborative Approach to Preventing and Treating Asthma in Infants and Young Children. January 2005. EJ847179
- [Background] Association AL. Asthma & Children Fact Sheet 2012. http://www.lung.org/lung-disease/asthma/resources/facts-and-figures/asthma-children-fact-sheet.html
- [Background] Farber HJ. Risk of readmission to hospital for pediatric asthma. J Asthma. 1998;35(1):95-9. doi: 10.3109/02770909809055410. PMID 9513588
- [Background] Minkovitz CS, Andrews JS, Serwint JR. Rehospitalization of children with asthma. Arch Pediatr Adolesc Med. 1999 Jul;153(7):727-30. doi: 10.1001/archpedi.153.7.727. PMID 10401806
- [Background] Lieu TA, Quesenberry CP, Sorel ME, Mendoza GR, Leong AB. Computer-based models to identify high-risk children with asthma. Am J Respir Crit Care Med. 1998 Apr;157(4 Pt 1):1173-80. doi: 10.1164/ajrccm.157.4.9708124. PMID 9563736
- [Background] Rea HH, Scragg R, Jackson R, Beaglehole R, Fenwick J, Sutherland DC. A case-control study of deaths from asthma. Thorax. 1986 Nov;41(11):833-9. doi: 10.1136/thx.41.11.833. PMID 3824270
- [Background] Weiss KB, Gergen PJ, Hodgson TA. An economic evaluation of asthma in the United States. N Engl J Med. 1992 Mar 26;326(13):862-6. doi: 10.1056/NEJM199203263261304. PMID 1542323
- [Background] Smith DH, Malone DC, Lawson KA, Okamoto LJ, Battista C, Saunders WB. A national estimate of the economic costs of asthma. Am J Respir Crit Care Med. 1997 Sep;156(3 Pt 1):787-93. doi: 10.1164/ajrccm.156.3.9611072. PMID 9309994
- [Background] Bloomberg GR, Trinkaus KM, Fisher EB Jr, Musick JR, Strunk RC. Hospital readmissions for childhood asthma: a 10-year metropolitan study. Am J Respir Crit Care Med. 2003 Apr 15;167(8):1068-76. doi: 10.1164/rccm.2201015. PMID 12684246
- [Background] Crane J, Pearce N, Burgess C, Woodman K, Robson B, Beasley R. Markers of risk of asthma death or readmission in the 12 months following a hospital admission for asthma. Int J Epidemiol. 1992 Aug;21(4):737-44. doi: 10.1093/ije/21.4.737. PMID 1521979
- [Background] Li D, German D, Lulla S, Thomas RG, Wilson SR. Prospective study of hospitalization for asthma. A preliminary risk factor model. Am J Respir Crit Care Med. 1995 Mar;151(3 Pt 1):647-55. doi: 10.1164/ajrccm.151.3.7881651.
- [Background] To T, Dick P, Feldman W, Hernandez R. A cohort study on childhood asthma admissions and readmissions. Pediatrics. 1996 Aug;98(2 Pt 1):191-5. PMID 8692616
- [Background] Chapman KR, Boulet LP, Rea RM, Franssen E. Suboptimal asthma control: prevalence, detection and consequences in general practice. Eur Respir J. 2008 Feb;31(2):320-5. doi: 10.1183/09031936.00039707. Epub 2007 Oct 24. PMID 17959642
- [Background] Centers for Disease Control and Prevention (CDC). Asthma hospitalizations and readmissions among children and young adults--Wisconsin, 1991-1995. MMWR Morb Mortal Wkly Rep. 1997 Aug 8;46(31):726-9. PMID 9262074
- [Background] Mitchell EA, Bland JM, Thompson JM. Risk factors for readmission to hospital for asthma in childhood. Thorax. 1994 Jan;49(1):33-6. doi: 10.1136/thx.49.1.33. PMID 8153938
- [Background] Vargas PA, Perry TT, Robles E, Jo CH, Simpson PM, Magee JM, Feild CR, Hakkak R, Carroll PA, Jones SM. Relationship of body mass index with asthma indicators in head start children. Ann Allergy Asthma Immunol. 2007 Jul;99(1):22-8. doi: 10.1016/S1081-1206(10)60616-3. PMID 17650825
- [Background] Barnes PJ. Achieving asthma control. Curr Med Res Opin. 2005;21 Suppl 4:S5-9. doi: 10.1185/030079905X61730. PMID 16138939
- [Background] Bloomberg GR, Banister C, Sterkel R, Epstein J, Bruns J, Swerczek L, Wells S, Yan Y, Garbutt JM. Socioeconomic, family, and pediatric practice factors that affect level of asthma control. Pediatrics. 2009 Mar;123(3):829-35. doi: 10.1542/peds.2008-0504. PMID 19255010
- [Background] Bateman ED, Frith LF, Braunstein GL. Achieving guideline-based asthma control: does the patient benefit? Eur Respir J. 2002 Sep;20(3):588-95. doi: 10.1183/09031936.02.00294702. PMID 12358333
- [Background] Rabe KF, Adachi M, Lai CK, Soriano JB, Vermeire PA, Weiss KB, Weiss ST. Worldwide severity and control of asthma in children and adults: the global asthma insights and reality surveys. J Allergy Clin Immunol. 2004 Jul;114(1):40-7. doi: 10.1016/j.jaci.2004.04.042. PMID 15241342
- [Background] National Asthma Education and Prevention Program. Expert Panel Report 3 (EPR-3): Guidelines for the Diagnosis and Management of Asthma-Summary Report 2007. J Allergy Clin Immunol. 2007 Nov;120(5 Suppl):S94-138. doi: 10.1016/j.jaci.2007.09.043. PMID 17983880
- [Background] Stempel DA, McLaughin TP, Stanford RH, Fuhlbrigge AL. Patterns of asthma control: a 3-year analysis of patient claims. J Allergy Clin Immunol. 2005 May;115(5):935-9. doi: 10.1016/j.jaci.2005.01.054. PMID 15867848
- [Background] Williams SG, Schmidt DK, Redd SC, Storms W; National Asthma Education and Prevention Program. Key clinical activities for quality asthma care. Recommendations of the National Asthma Education and Prevention Program. MMWR Recomm Rep. 2003 Mar 28;52(RR-6):1-8. PMID 12696781
- [Background] New NHLBI guidelines for the diagnosis and management of asthma. National Heart, Lung and Blood Institute. Lippincott Health Promot Lett. 1997 Aug;2(7):1, 8-9. No abstract available. PMID 9300898
- [Background] Glauber JH, Farber HJ, Homer CJ. Asthma clinical pathways: toward what end? Pediatrics. 2001 Mar;107(3):590-2. doi: 10.1542/peds.107.3.590. No abstract available. PMID 11230605
- [Background] Ressel GW; Centers for Disease Control and Prevention; National Asthma Education and Prevention Program. NAEPP updates guidelines for the diagnosis and management of asthma. Am Fam Physician. 2003 Jul 1;68(1):169-70. No abstract available. PMID 12887123
- [Background] Jovicic A, Holroyd-Leduc JM, Straus SE. Effects of self-management intervention on health outcomes of patients with heart failure: a systematic review of randomized controlled trials. BMC Cardiovasc Disord. 2006 Nov 2;6:43. doi: 10.1186/1471-2261-6-43. PMID 17081306
- [Background] Clark DO, Frankel RM, Morgan DL, Ricketts G, Bair MJ, Nyland KA, Callahan CM. The meaning and significance of self-management among socioeconomically vulnerable older adults. J Gerontol B Psychol Sci Soc Sci. 2008 Sep;63(5):S312-9. doi: 10.1093/geronb/63.5.s312. PMID 18818452
- [Background] McGowan P. Self-Managment: A Background Paper. Centre on Aging New Perspectives: International Conference on Patient Self-Management 2006:1-10.
- [Background] Barlow J, Wright C, Sheasby J, Turner A, Hainsworth J. Self-management approaches for people with chronic conditions: a review. Patient Educ Couns. 2002 Oct-Nov;48(2):177-87. doi: 10.1016/s0738-3991(02)00032-0. PMID 12401421
- [Background] Adams WG, Fuhlbrigge AL, Miller CW, Panek CG, Gi Y, Loane KC, Madden NE, Plunkett AM, Friedman RH. TLC-Asthma: an integrated information system for patient-centered monitoring, case management, and point-of-care decision support. AMIA Annu Symp Proc. 2003;2003:1-5. PMID 14728122
- [Background] Cruz-Correia R, Fonseca J, Lima L, Araujo L, Delgado L, Castel-Branco MG, Costa-Pereira A. Web-based or paper-based self-management tools for asthma--patients' opinions and quality of data in a randomized crossover study. Stud Health Technol Inform. 2007;127:178-89. PMID 17901611
- [Background] Finkelstein J, Cabrera MR, Hripcsak G. Internet-based home asthma telemonitoring: can patients handle the technology? Chest. 2000 Jan;117(1):148-55. doi: 10.1378/chest.117.1.148. PMID 10631213
- [Background] Janson SL, McGrath KW, Covington JK, Cheng SC, Boushey HA. Individualized asthma self-management improves medication adherence and markers of asthma control. J Allergy Clin Immunol. 2009 Apr;123(4):840-6. doi: 10.1016/j.jaci.2009.01.053. PMID 19348923
- [Background] Joshi A, Amelung P, Arora M, Finkelstein J. Clinical impact of home automated telemanagement in asthma. AMIA Annu Symp Proc. 2005;2005:1000. PMID 16779287
- [Background] Ostojic V, Cvoriscec B, Ostojic SB, Reznikoff D, Stipic-Markovic A, Tudjman Z. Improving asthma control through telemedicine: a study of short-message service. Telemed J E Health. 2005 Feb;11(1):28-35. doi: 10.1089/tmj.2005.11.28. PMID 15785218
- [Background] van der Meer V, van Stel HF, Bakker MJ, Roldaan AC, Assendelft WJ, Sterk PJ, Rabe KF, Sont JK; SMASHING (Self-Management of Asthma Supported by Hospitals, ICT, Nurses and General practitioners) Study Group. Weekly self-monitoring and treatment adjustment benefit patients with partly controlled and uncontrolled asthma: an analysis of the SMASHING study. Respir Res. 2010 Jun 10;11(1):74. doi: 10.1186/1465-9921-11-74. PMID 20537124
- [Background] Ahmad E, Grimes DE. The effects of self-management education for school-age children on asthma morbidity: a systematic review. J Sch Nurs. 2011 Aug;27(4):282-92. doi: 10.1177/1059840511403003. Epub 2011 Apr 8. PMID 21478414
- [Background] Bonner S, Zimmerman BJ, Evans D, Irigoyen M, Resnick D, Mellins RB. An individualized intervention to improve asthma management among urban Latino and African-American families. J Asthma. 2002 Apr;39(2):167-79. doi: 10.1081/jas-120002198. PMID 11990232
- [Background] Perneger TV, Sudre P, Muntner P, Uldry C, Courteheuse C, Naef AF, Jacquemet S, Nicod L, Rochat T, Assal JP. Effect of patient education on self-management skills and health status in patients with asthma: a randomized trial. Am J Med. 2002 Jul;113(1):7-14. doi: 10.1016/s0002-9343(02)01136-1. PMID 12106617
- [Background] Rhee H, Belyea MJ, Hunt JF, Brasch J. Effects of a peer-led asthma self-management program for adolescents. Arch Pediatr Adolesc Med. 2011 Jun;165(6):513-9. doi: 10.1001/archpediatrics.2011.79. PMID 21646583
- [Background] Guendelman S, Meade K, Benson M, Chen YQ, Samuels S. Improving asthma outcomes and self-management behaviors of inner-city children: a randomized trial of the Health Buddy interactive device and an asthma diary. Arch Pediatr Adolesc Med. 2002 Feb;156(2):114-20. doi: 10.1001/archpedi.156.2.114. PMID 11814370
- [Background] Bheekie A, Syce JA, Weinberg EG. Peak expiratory flow rate and symptom self-monitoring of asthma initiated from community pharmacies. J Clin Pharm Ther. 2001 Aug;26(4):287-96. doi: 10.1046/j.1365-2710.2001.00361.x. PMID 11493372
- [Background] Thompson R, Delfino RJ, Tjoa T, Nussbaum E, Cooper D. Evaluation of daily home spirometry for school children with asthma: new insights. Pediatr Pulmonol. 2006 Sep;41(9):819-28. doi: 10.1002/ppul.20449. PMID 16847876
- [Background] Chan DS, Callahan CW, Hatch-Pigott VB, Lawless A, Proffitt HL, Manning NE, Schweikert M, Malone FJ. Internet-based home monitoring and education of children with asthma is comparable to ideal office-based care: results of a 1-year asthma in-home monitoring trial. Pediatrics. 2007 Mar;119(3):569-78. doi: 10.1542/peds.2006-1884. PMID 17332210
- [Background] de Jongste JC, Carraro S, Hop WC; CHARISM Study Group; Baraldi E. Daily telemonitoring of exhaled nitric oxide and symptoms in the treatment of childhood asthma. Am J Respir Crit Care Med. 2009 Jan 15;179(2):93-7. doi: 10.1164/rccm.200807-1010OC. Epub 2008 Oct 17. PMID 18931330
- [Background] McPherson AC, Glazebrook C, Forster D, James C, Smyth A. A randomized, controlled trial of an interactive educational computer package for children with asthma. Pediatrics. 2006 Apr;117(4):1046-54. doi: 10.1542/peds.2005-0666. PMID 16585298
- [Background] Willems DC, Joore MA, Hendriks JJ, Nieman FH, Severens JL, Wouters EF. The effectiveness of nurse-led telemonitoring of asthma: results of a randomized controlled trial. J Eval Clin Pract. 2008 Aug;14(4):600-9. doi: 10.1111/j.1365-2753.2007.00936.x. Epub 2008 Jul 9. PMID 19126178
- [Background] Jan RL, Wang JY, Huang MC, Tseng SM, Su HJ, Liu LF. An internet-based interactive telemonitoring system for improving childhood asthma outcomes in Taiwan. Telemed J E Health. 2007 Jun;13(3):257-68. doi: 10.1089/tmj.2006.0053. PMID 17603828
- [Background] Joseph CL, Peterson E, Havstad S, Johnson CC, Hoerauf S, Stringer S, Gibson-Scipio W, Ownby DR, Elston-Lafata J, Pallonen U, Strecher V; Asthma in Adolescents Research Team. A web-based, tailored asthma management program for urban African-American high school students. Am J Respir Crit Care Med. 2007 May 1;175(9):888-95. doi: 10.1164/rccm.200608-1244OC. Epub 2007 Feb 8. PMID 17290041
- [Background] NHLBI. So You Have Asthma. 2007(NIH Publication No. 07-5248). https://www.nhlbi.nih.gov/files/docs/public/lung/have_asthma.pdf.
- [Background] Cuijpers CE, Wesseling GJ, Swaen GM, Sturmans F, Wouters EF. Asthma-related symptoms and lung function in primary school children. J Asthma. 1994;31(4):301-12. doi: 10.3109/02770909409089477. PMID 8040154
- [Background] Davis KJ, Disantostefano R, Peden DB. Is Johnny wheezing? Parent-child agreement in the Childhood Asthma in America survey. Pediatr Allergy Immunol. 2011 Feb;22(1 Pt 1):31-5. doi: 10.1111/j.1399-3038.2010.01016.x. Epub 2010 Sep 9. PMID 21261742
- [Background] Halterman JS, Yoos HL, Kitzman H, Anson E, Sidora-Arcoleo K, McMullen A. Symptom reporting in childhood asthma: a comparison of assessment methods. Arch Dis Child. 2006 Sep;91(9):766-70. doi: 10.1136/adc.2006.096123. Epub 2006 May 16. PMID 16705016
- [Background] McQuaid EL, Koinis Mitchell D, Walders N, Nassau JH, Kopel SJ, Klein RB, Wamboldt MZ, Fritz GK. Pediatric asthma morbidity: the importance of symptom perception and family response to symptoms. J Pediatr Psychol. 2007 Mar;32(2):167-77. doi: 10.1093/jpepsy/jsj112. Epub 2006 May 22. PMID 16717140
- [Background] Hagmolen Of Ten Have W, van den Berg NJ, van der Palen J, van Aalderen WM, Bindels PJ. Limitations of questioning asthma to assess asthma control in general practice. Respir Med. 2008 Aug;102(8):1153-8. doi: 10.1016/j.rmed.2008.03.008. Epub 2008 Jun 24. PMID 18573649
- [Background] Bridge PD, McKenzie SA. Bronchodilator responsiveness testing in young children. Arch Dis Child. 2001 Jun;84(6):525. doi: 10.1136/adc.84.6.525n. No abstract available. PMID 11372088
- [Background] NHLBI-EPR-3. Guidelines for the diagnosis ane management of asthma. Periodic Assessment and Monitoring: Essential for Asthma Management. 2007. http://www.nhlbi.nih.gov/files/docs/guidelines/asthsumm.pdf
- [Background] Tirimanna PR, Den Otter JJ, Van Schayck CP, Van Herwaarden CL, Folgering H, Van Weel C. Evaluation of the suitability of weekly peak expiratory flow rate measurements in monitoring annual decline in lung function among patients with asthma and chronic bronchitis. Br J Gen Pract. 1996 Jan;46(402):15-8. PMID 8745846
- [Background] Frischer T, Meinert R, Urbanek R, Kuehr J. Variability of peak expiratory flow rate in children: short and long term reproducibility. Thorax. 1995 Jan;50(1):35-9. doi: 10.1136/thx.50.1.35. PMID 7886646
- [Background] Goldberg S, Springer C, Avital A, Godfrey S, Bar-Yishay E. Can peak expiratory flow measurements estimate small airway function in asthmatic children? Chest. 2001 Aug;120(2):482-8. doi: 10.1378/chest.120.2.482. PMID 11502647
- [Background] Liu AH, Zeiger R, Sorkness C, Mahr T, Ostrom N, Burgess S, Rosenzweig JC, Manjunath R. Development and cross-sectional validation of the Childhood Asthma Control Test. J Allergy Clin Immunol. 2007 Apr;119(4):817-25. doi: 10.1016/j.jaci.2006.12.662. Epub 2007 Mar 13. PMID 17353040
- [Background] Nathan RA, Sorkness CA, Kosinski M, Schatz M, Li JT, Marcus P, Murray JJ, Pendergraft TB. Development of the asthma control test: a survey for assessing asthma control. J Allergy Clin Immunol. 2004 Jan;113(1):59-65. doi: 10.1016/j.jaci.2003.09.008. PMID 14713908
- [Background] McGrath AM, Gardner DM, McCormack J. Is home peak expiratory flow monitoring effective for controlling asthma symptoms? J Clin Pharm Ther. 2001 Oct;26(5):311-7. doi: 10.1046/j.1365-2710.2001.00374.x. PMID 11679021
- [Background] Juniper EF, Gruffydd-Jones K, Ward S, Svensson K. Asthma Control Questionnaire in children: validation, measurement properties, interpretation. Eur Respir J. 2010 Dec;36(6):1410-6. doi: 10.1183/09031936.00117509. Epub 2010 Jun 7. PMID 20530041
- [Background] Kattan M. Quality of inpatient care for asthma: challenges and opportunities. Pediatrics. 2008 Dec;122(6):1369-70. doi: 10.1542/peds.2008-2787. No abstract available. PMID 19047258

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard e-Asthma Tracker (e-AT) Intervention: Patients in Standard e-AT intervention group will be using the standard version of e-AT
- Intensive e-Asthma Tracker (e-AT) Intervention: Participants in the intensive e-AT intervention group will be using an enhanced version of the standard e-AT, i.e. addition of progress bar indicating the patients' status of completing 4 scores in a month, fireworks when they reach 100% on the progress bar, a leaderboard to compare their own status among other e-AT users.
Period: Overall Study
Arm/Group | Standard e-Asthma Tracker (e-AT) Intervention | Intensive e-Asthma Tracker (e-AT) Intervention | Usual Care (Non-Randomized Cohort)
Started | 267 | 60 | 599
3 Months Follow-up | 178 | 40 | 599
6 Months Follow-up | 182 | 42 | 599
12 Months Follow-up | 167 | 43 | 599
Completed | 167 | 43 | 599
Not Completed | 100 | 17 | 0

BASELINE CHARACTERISTICS:
Groups:
- Standard e-AT Intervention: Patients in Standard e-AT intervention group will be using the standard version of e-AT.
- Intensive e-AT Intervention: Participants in the intensive e-AT intervention group will be using an enhanced version of the standard e-AT, i.e. addition of progress bar indicating the patients' status of completing 4 scores in a month, fireworks when they reach 100% on the progress bar, a leaderboard to compare their own status among other e-AT users.
- Total: Total of all reporting groups
Arm/Group | Standard e-AT Intervention | Intensive e-AT Intervention | Usual Care (Non-Randomized Cohort) | Total
Number analyzed (Participants) | 267 | 60 | 599 | 926
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 267 | 60 | 599 | 926
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.12 (3.99) | 7.18 (8.12) | 8.04 (3.86) | 7.97 (3.89)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 110 | 23 | 228 | 361
  Male | 157 | 37 | 371 | 565
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 40 | 4 | 72 | 116
  Not Hispanic or Latino | 216 | 53 | 520 | 789
  Unknown or Not Reported | 11 | 3 | 7 | 21
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 5 | 1 | 5 | 11
  Asian | 3 | 1 | 11 | 15
  Native Hawaiian or Other Pacific Islander | 7 | 0 | 9 | 16
  Black or African American | 9 | 1 | 23 | 33
  White | 223 | 51 | 537 | 811
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 20 | 6 | 14 | 40
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 267 | 60 | 599 | 926

OUTCOME MEASURES:

1. Primary Outcome: Patient Quality of Life (QOL), Compared Mean QOL Change From Baseline at Each Follow-up Assessment Between the Clinics Assigned to the Intensive and Standard e-AT Interventions
Description: Patient QOL and missed school days was collected longitudinally through surveys of the study population defined above. The QOL questionnaire included the Integrated Therapeutics Group Child Asthma Short Form (ITG-CASF) and was used at baseline (at first assessment), 3, 6, and 12 months in the study.
  Items within QOL scales are summed and linearly transformed from 0 to 100, with higher scores indicating better functioning.
Time Frame: Quality of Life assessed at baseline, then compared to 3 months, 6 months, and 12 months after intervention.
Population: We enrolled 327, 2 clinics with only 1 patient enrolled were excluded, leaving 325 patients. Of 325, 7 did not provide baselines and were excluded, leaving 318 (261 standard vs. 57 intensive) participants. Row numbers differ due to different number of participants completing 3, 6, and 12 months follow-ups, due to withdrawal and loss to follow-up.
Measure: Mean (Standard Error); unit: Units on a scale
Groups:
- Standard e-AT Intervention: Patients in Standard e-AT intervention group using the standard version of e-AT.
- Intensive e-AT Intervention: Participants in the intensive e-AT intervention group using an enhanced version of the standard e-AT, i.e. addition of progress bar indicating the patients' status of completing 4 scores in a month, fireworks when they reach 100% on the progress bar, a leaderboard to compare their own status among other e-AT users.
Arm/Group | Standard e-AT Intervention | Intensive e-AT Intervention
Number analyzed (Participants) | 261 | 57
Units on a scale
  3 Months Follow-up vs Baseline: number analyzed (Participants) | 178 | 40
  3 Months Follow-up vs Baseline | 8.55 (0.97) | 7.64 (2.53)
  6 Months Follow-up compared vs Baseline: number analyzed (Participants) | 182 | 42
  6 Months Follow-up compared vs Baseline | 8.37 (0.86) | 5.78 (1.94)
  12 Months Follow-up vs Baseline: number analyzed (Participants) | 167 | 43
  12 Months Follow-up vs Baseline | 9.39 (0.76) | 9.29 (1.80)

2. Primary Outcome: Patient Quality of Life (QOL), Overall Longitudinal Change (From Baseline) Within All Subjects (Who Received the e-AT Intervention)
Description: Patient QOL and missed school days was collected longitudinally through surveys of the study population defined above. The QOL questionnaire included the Integrated Therapeutics Group Child Asthma Short Form - ITG-CASF and was used at baseline (at first assessment), 3, 6, and 12 months in the study. Items within scales are summed and linearly transformed from 0 to 100, with higher scores indicating better functioning.
Time Frame: Average Baseline QOL was compared to QOL scores at 3, 6 and 12 month follow-up QOL
Population: The numbers analyzed in the rows are different due to different number of participants completing the surveys throughout 3, 6, and 12 months. This was due to withdrawal from the study or loss to follow-up.
Measure: Mean (Standard Deviation); unit: units (points) on a scale, range 0-100
Groups:
- All e-AT Users: This group consists of all e-AT users, both standard and intensive interventions.
Arm/Group | All e-AT Users
Number analyzed (Participants) | 318
units (points) on a scale, range 0-100
  Baseline | 79.07 (14.20)
  3 Months: number analyzed (Participants) | 218
  3 Months | 90.98 (9.54)
  6 Months: number analyzed (Participants) | 224
  6 Months | 90.04 (11.12)
  12 Months: number analyzed (Participants) | 210
  12 Months | 90.64 (10.34)

3. Secondary Outcome: Parent Satisfaction With Care, Standard vs Intensive
Description: Parent satisfaction data was collected at baseline and at 12 months in the study.
  The scale ranges from 1-5, with 1 being "Very Dissatisfied" and 5 "Very Satisfied".
Time Frame: Changes in satisfaction was compared between 12 month follow-up and baseline satisfaction across Standard and Intensive interventions
Population: We had 261 in Standard e-AT and 57 in Intensive e-AT who completed baseline survey, and 166 in Standard e-AT and 42 in Intensive e-AT completed the 12 Months Follow-up Survey. This is due to participant withdrawal and loss to follow-up.
Measure: Mean (95% Confidence Interval); unit: units (points) on a scale (from 1-5)
Arm/Group | Standard e-AT Intervention | Intensive e-AT Intervention
Number analyzed (Participants) | 261 | 57
units (points) on a scale (from 1-5)
  Baseline | 4.63 [4.49 to 4.77] | 4.63 [4.49 to 4.77]
  12 months Follow-up: number analyzed (Participants) | 166 | 42
  12 months Follow-up | 4.38 [4.23 to 4.53] | 4.54 [4.35 to 4.72]

4. Secondary Outcome: Child Interrupted/Missed School Days, Standard vs Intensive
Description: Number of child interrupted/missed school days were collected longitudinally at the same time as collecting the QOL scores: baseline, 3, 6, and 12 months in the study.
  Number of child interrupted/missed school days during the 3 months prior to baseline, 3, 6, and 12 months follow-up surveys were counted.
Time Frame: Interrupted/missed school days were collected at baseline, 3, 6, and 12 month follow-ups
Population: We had 261 Standard and 57 Intensive e-AT who completed baseline survey. Numbers in the row differ due to different number of participants who completed 3, 6, and 12 months surveys, due to participant compliance, withdrawal or loss-to-follow-up. 3, 6, and 12 month measurements were compared to Baseline, between Standard vs Intensive interventions
Measure: Number; unit: Number of interrupted/missed school days
Arm/Group | Standard e-AT Intervention | Intensive e-AT Intervention
Number analyzed (Participants) | 261 | 57
Number of interrupted/missed school days
  Baseline | 435 | 129
  3 Months Follow-up: number analyzed (Participants) | 178 | 40
  3 Months Follow-up | 114 | 60
  6 Months Follow-up: number analyzed (Participants) | 182 | 42
  6 Months Follow-up | 87 | 30
  12 Months Follow-up: number analyzed (Participants) | 167 | 43
  12 Months Follow-up | 129 | 37

5. Secondary Outcome: Parent Interrupted/Missed Work Days, Standard vs Intensive
Description: Number of parent interrupted/missed work days were collected longitudinally at the same time as collecting the QOL scores: baseline, 3, 6, and 12 months in the study.
  Number of parent interrupted/missed work days during the 3 months prior to baseline, 3, 6, and 12 months follow-up surveys were counted.
Time Frame: Interrupted/missed work days were measured baseline 3, 6, and 12 months
Population: as for outcome 4
Measure: Number; unit: Number of interrupted/missed work days
Arm/Group | Standard e-AT Intervention | Intensive e-AT Intervention
Number analyzed (Participants) | 261 | 57
Number of interrupted/missed work days
  Baseline | 176 | 56
  3 Months Follow-up: number analyzed (Participants) | 178 | 40
  3 Months Follow-up | 44 | 14
  6 Months Follow-up: number analyzed (Participants) | 182 | 42
  6 Months Follow-up | 42 | 15
  12 Months Follow-up: number analyzed (Participants) | 167 | 43
  12 Months Follow-up | 23 | 18

6. Secondary Outcome: Asthma Control Change, Standard vs Intensive
Description: Asthma control information was collected weekly through the e-AT for 1 year. Asthma control was measured using the Asthma Control Test (ACT), which had a score ranging from 5 to 25, with 5 being poor control and 25 being optimal control. The analysis compared the mean change in scores from baseline to quarters 1, 2, 3, and 4.
Time Frame: Average baseline ACT scores compared to average ACT scores at quarter 1, 2, 3 and 4, and between Standard vs. Intensive
Measure: Mean (Standard Error); unit: mean score (points) change
Arm/Group | Standard e-AT Intervention | Intensive e-AT Intervention
Number analyzed (Participants) | 261 | 57
mean score (points) change
  Qtr 1 vs baseline | 2.55 (0.12) | 1.78 (0.35)
  Qtr 2 vs baseline | 3.09 (0.10) | 2.18 (0.30)
  Qtr 3 vs baseline | 3.26 (0.09) | 2.18 (0.23)
  Qtr 4 vs baseline | 3.33 (0.10) | 3.30 (0.22)

7. Secondary Outcome: Emergency Department (ED)/Hospitalization, Standard vs Intensive
Description: ED and hospital admissions were evaluated using data collected through Intermountain Healthcare claims data and ED visits and hospital encounters.
  We evaluated number ED and hospital admissions 12 months prior to intervention and 12 months post intervention
Time Frame: Change in 1 year ED/hospital admission between 12-month prior and 12 month post e-AT use
Population: Number of pre- and post e-AT ED and hospital admissions were compared between standard and intensive groups.
Measure: Number; unit: Number of ED/hospital admissions
Arm/Group | Standard e-AT Intervention | Intensive e-AT Intervention
Number analyzed (Participants) | 261 | 57
Number of ED/hospital admissions
  Prior | 53 | 18
  Post | 21 | 8

8. Secondary Outcome: Parent Satisfaction With Care, Overall (Change Overtime From Baseline to 12 Months)
Description: Parent satisfaction data was collected using a modified version of patient satisfaction survey developed and validated by Varni et al. at baseline and at 12 months in the study.
  The scale ranged from 1-5, with 1=Very Dissatisfied and 5=Very Satisfied.
Time Frame: Satisfaction at 1 year following e-AT use was compared to baseline satisfaction scores
Population: We had 318 participants who have completed the baseline satisfaction survey, and 208 who completed 12 months follow-up survey, due to participants withdrawing from the study and loss to follow-up.
Measure: Mean (Standard Deviation); unit: units (points) on a scale (from 1-5)
Arm/Group | All e-AT Users
Number analyzed (Participants) | 318
units (points) on a scale (from 1-5)
  Baseline | 4.66 (0.51)
  12 months Follow-up: number analyzed (Participants) | 208
  12 months Follow-up | 4.46 (0.53)

9. Secondary Outcome: Child Asthma Control Overall (Comparing Change of Asthma Control From Baseline to Quarter 1, Quarter 2, Quarter 3 and Quarter 4)
Description: Asthma control information was collected through the e-AT, comparing change of asthma control from baseline to quarter 1, quarter 2, quarter 3 and quarter 4.
  Asthma control was measured using the Asthma Control Test (ACT), which scale ranged from 5-25, with 5=poorly controlled and 25=well controlled.
  Each patient submitted an ACT score weekly for 12 months.
Time Frame: baseline ACT scores were compared to quarters 1, 2, 3, 4.
Population: Patients were told to submit an ACT score once a week for 12 months. 311 patients completed at least one ACT score for a total number of 11418 ACT scores submitted using e-AT by all e-AT users (during study period).
Measure: Mean (Standard Deviation); unit: Score (points) ranging from 5-25
Units Other Than Participants: ACT scores
Groups:
- All e-AT Users: This group consists of all e-AT users, both standard and intensive interventions. We will be looking at ACT scores submitted by the e-AT users to report asthma control over 12 months.
Arm/Group | All e-AT Users
Number analyzed (Participants) | 311
Number analyzed (ACT scores) | 11418
Score (points) ranging from 5-25
  Baseline: number analyzed (ACT scores) | 311
  Baseline | 18.85 (5.49)
  Quarter 1: number analyzed (ACT scores) | 2965
  Quarter 1 | 22.28 (3.25)
  Quarter 2: number analyzed (ACT scores) | 2861
  Quarter 2 | 22.82 (2.95)
  Quarter 3: number analyzed (ACT scores) | 2726
  Quarter 3 | 22.81 (2.98)
  Quarter 4: number analyzed (ACT scores) | 2555
  Quarter 4 | 22.97 (2.76)

10. Secondary Outcome: Child Interrupted/Missed School Days, Overall (Longitudinal Changes Overtime)
Description: Number of child interrupted/missed school days were collected longitudinally (information includes mean at baseline, 3, 6, and 12 months in the study).
Time Frame: 1 year
Population: The numbers analyzed in the rows are different due to different number of participants completing the surveys throughout 3, 6, and 12 months. This was due to either compliance, withdrawal or loss to follow-up.
Measure: Mean (Standard Deviation); unit: Number of days (interrupted or missed)
Arm/Group | All e-AT Users
Number analyzed (Participants) | 318
Number of days (interrupted or missed)
  Baseline | 1.91 (5.18)
  3 Months Follow-up: number analyzed (Participants) | 218
  3 Months Follow-up | 0.80 (2.07)
  6 Months Follow-up: number analyzed (Participants) | 224
  6 Months Follow-up | 0.52 (1.34)
  12 Months Follow-up: number analyzed (Participants) | 210
  12 Months Follow-up | 0.79 (2.06)

11. Secondary Outcome: Parent Interrupted/Missed Work Days, Overall (Longitudinal Change Overtime)
Description: Number of parent interrupted/missed work days were collected longitudinally at the same time as collecting the QOL scores: Information includes mean at baseline, 3, 6, and 12 months in the study.
Time Frame: 1 year
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Number of days (interrupted or missed)
Arm/Group | All e-AT Users
Number analyzed (Participants) | 318
Number of days (interrupted or missed)
  Baseline | 0.72 (1.89)
  3 Months Follow-up: number analyzed (Participants) | 218
  3 Months Follow-up | 0.27 (0.99)
  6 Months Follow-Up: number analyzed (Participants) | 224
  6 Months Follow-Up | 0.25 (1.02)
  12 Months Follow-up: number analyzed (Participants) | 210
  12 Months Follow-up | 0.20 (0.83)

12. Secondary Outcome: ED/Hospital Admissions, e-AT Overall (Pre vs. Post e-AT Use Within Subjects That Received the e-AT Intervention)
Description: ED/hospital re-admission data were compared between prior and post 12 month period (for both intensive and standard interventions overall) when e-AT was administered.
Time Frame: 1 year
Population: Here we used intent-to-treat analysis and included the overall 325 (rather than 318 used in analysis of other outcomes) participants
Measure: Mean (Standard Deviation); unit: number of ED/hospital admission
Groups:
- Prior e-AT Use: The participants enrolled in both standard and intensive e-AT groups served as their own control. This arm includes ED/Hospital use among the participants 1 year before using the e-AT.
- Post e-AT Use: The participants enrolled in both standard and intensive e-AT groups served as their own control. This arm includes ED/Hospital use among the participants 1 year after starting using the e-AT.
Arm/Group | Prior e-AT Use | Post e-AT Use
Number analyzed (Participants) | 325 | 325
number of ED/hospital admission | 0.22 (0.60) | 0.09 (0.35)

13. Secondary Outcome: Use of Oral Steroid, Overall
Description: Use of oral steroid was evaluated using data collected through Intermountain Healthcare claims data and oral steroids prescribed. Comparison was made between prior and post e-AT (both interventions) overall.
Time Frame: 1 year
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: number of oral steroid use
Groups:
- Prior e-AT Use: The participants enrolled in both standard and intensive e-AT groups served as their own control. This arm includes oral steriod use among the participants 1 year before using the e-AT.
- Post e-AT Use: The participants enrolled in both standard and intensive e-AT groups served as their own control. This arm includes the oral steriod use among the participants 1 year after starting using the e-AT.
Arm/Group | Prior e-AT Use | Post e-AT Use
Number analyzed (Participants) | 325 | 325
number of oral steroid use | 0.74 (1.15) | 0.51 (0.95)

14. Secondary Outcome: ED/Hospital Admission, Early vs. Late Patients
Description: ED and hospital admission was evaluated using data collected through Intermountain Healthcare claims data and ED visits and hospital encounters. Analyses (at the patient level) comparing the rates of ED/hospital admissions between a 1 year period following initiation of the e-AT for those in both standard and intensive e-AT groups who were enrolled early during the study period (patients with enrollment dates between January 2014 and December 2014) to rates of ED/hospital admissions for patients who started the e-AT later (patients with enrollment dates between January 2015 and December 2015), during a 1-year period prior to the late patient starting the e-AT.
Time Frame: 1 year following e-AT use for early and late starting patients
Population: Intent-to-treat analysis was used, including all 325. Randomized comparisons compared intensive vs. standard e-AT, but not e-AT efficacy vs usual care. This nonrandomized analysis (Early vs Late Patients) assesses e-AT efficacy, comparing outcomes between "period" patients were under the e-AT vs "periods" other patients were not using the e-AT.
Measure: Mean (Standard Deviation); unit: number of ED/Hospital admission
Groups:
- Early Starting Patients: Patients starting with e-AT intervention early (in 2014)
- Late Starting Patients: Patients starting with e-AT intervention later (in 2015)
Arm/Group | Early Starting Patients | Late Starting Patients
Number analyzed (Participants) | 234 | 91
number of ED/Hospital admission | 0.10 (0.38) | 0.18 (0.10)

15. Secondary Outcome: Oral Steroid Use, Early vs. Late Patients
Description: Oral steroid use data was collected through Intermountain Healthcare claims data and clinics prescribing oral steroid.
  Oral steroid use was evaluated using data collected through Intermountain Healthcare claims data and oral steroids prescribed. Analyses (at the patient level) comparing the rates oral steroid use between a 1 year period following initiation of the e-AT for those in both standard and intensive e-AT groups who were enrolled early during the study period (patients with enrollment dates between January 2014 and December 2014) to rates of oral steroid use for patients who started the e-AT later (patients with enrollment dates between January 2015 and December 2015), during a 1-year period prior to the late patient starting the e-AT.
Time Frame: 1 year
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: number of oral steroid use
Arm/Group | Early Starting Patients | Late Starting Patients
Number analyzed (Participants) | 234 | 91
number of oral steroid use | 0.53 (0.99) | 0.53 (0.92)

16. Secondary Outcome: ED/Hospital Admission, Early vs Late Starting Clinics (During the 3 Months When Late Starting Clinics Have Not Used the e-AT)
Description: ED and hospital admission evaluated using data collected through Intermountain Healthcare claims data and ED visits and hospital encounters. Statistical analysis was not conducted since the numbers of ED/Hospital admissions was very small (2 and 0) in both group (during the 3 months study window). Here we used intent-to-treat analysis and included the overall 325 (rather than 318 used in analysis of other outcomes) participants.
Time Frame: 3-month period prior to the late clinics starting the e-AT
Population: Intent-to-treat analysis was used, including all 325. Randomized comparisons compared intensive vs. standard e-AT, but not e-AT efficacy vs usual care. This nonrandomized analysis (Early vs Late Clinics) assesses e-AT efficacy, comparing outcomes between "period" clinics were under the e-AT vs "periods" other clinics were not using the e-AT.
Measure: Number; unit: number of ED/Hospital admission
Groups:
- Early Starting Clinics: ED/Hospital admission for patients in clinics that started with the e-AT intervention from Jan 3, 2014 to Mar 24, 2014.
- Late Starting Clinics: ED/Hospital admission for patients in clinics that started with the e-AT intervention after March 24, 2014.
Arm/Group | Early Starting Clinics | Late Starting Clinics
Number analyzed (Participants) | 206 | 119
number of ED/Hospital admission | 2 | 0

17. Secondary Outcome: Oral Steroid Use, Early vs Late Starting Clinics (During the 3 Months When Late Starting Clinics Have Not Started the e-AT)
Description: Use of oral steroid was evaluated using data collected through Intermountain Healthcare claims data and oral steroids prescribed. Statistical analysis was not conducted since the numbers of ED/Hospital admissions was very small (2 and 0) in both group (during the 3 months study window). Here we used intent-to-treat analysis and included the overall 325 (rather than 318 used in analysis of other outcomes) participants
Time Frame: 3 month period prior to the late clinics starting the e-AT
Population: as for outcome 16
Measure: Number; unit: number of oral steroid use
Groups:
- Early Patients: Oral steroid use between Jan 3, 2014-March 24, 2014 for patients who were enrolled in e-AT intervention from Jan 3, 2014 to Mar 24, 2014.
- Late Patients: Oral steroid use between Jan 3, 2014-March 24, 2014 for patients who were enrolled into e-AT after March 24, 2014.
Arm/Group | Early Patients | Late Patients
Number analyzed (Participants) | 206 | 119
number of oral steroid use | 4 | 0

18. Secondary Outcome: ED/Hospital Admissions, e-AT vs Usual Care
Description: Non randomized comparison of ED and hospital admissions between e-AT interventions (both intensive and standard) compared usual care (matched control patients drawn from non-participating clinics) in the prior vs. post e-AT intervention time periods.
Time Frame: 1 year
Population: Here we used intent-to-treat analysis and included the overall 325 (rather than 318 used in analysis of other outcomes) e-AT participants and 599 matched controls retrieved electronically from non-participating clinics.
Measure: Mean (Standard Deviation); unit: Rate per 1000-days
Groups:
- e-AT Intervention: All e-AT users who have received the e-AT intervention for 12 months, randomized to either standard or intensive group.
- Usual Care (Non-randomized Cohort): Those who have not received any e-AT intervention and received usual care.
Arm/Group | e-AT Intervention | Usual Care (Non-randomized Cohort)
Number analyzed (Participants) | 325 | 599
Rate per 1000-days
  Prior | 0.59 (1.64) | 0.23 (1.01)
  Post | 0.24 (0.97) | 0.24 (0.97)

19. Secondary Outcome: Oral Steroid Use, e-AT vs Usual Care
Description: Non randomized comparison of use of oral steroid between e-AT interventions (both intensive and standard) compared usual care (matched control patients drawn from non-participating clinics) in the prior vs. post e-AT intervention time periods.
Time Frame: 1 year
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: Rate per 1000-days
Groups:
- Usual Care (Non-randomized Cohort): Matched control participants from non-participating clinics that have not received any e-AT intervention and received usual care.
Arm/Group | e-AT Intervention | Usual Care (Non-randomized Cohort)
Number analyzed (Participants) | 325 | 599
Rate per 1000-days
  Prior | 2.02 (3.14) | 1.87 (3.12)
  Post | 1.41 (2.60) | 1.99 (7.89)

ADVERSE EVENTS:
Description: This study is a minimal risk study, with patients logging in to a secure web-based self-management tool and answering questions about their asthma symptoms. The only intervention in the study was to have patients use this tool to manage asthma. No serious adverse risk is involved in this study.
Arm/Group | Standard e-AT Intervention | Intensive e-AT Intervention | Usual Care (Non-Randomized Cohort)
Serious Adverse Events (participants affected / at risk) | 0/267 | 0/60 | 0/599
Other Adverse Events (participants affected / at risk) | 0/267 | 0/60 | 0/599

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No